CLINICAL TRIAL: NCT05504070
Title: Venclose digiRF System: A Post-Market, Multi-Center, Prospective, Interventional Study for Treatment of Chronic Venous Disease of the Great and Small Saphenous Veins and Incompetent Perforator Veins
Brief Title: Venclose digiRF System Post Market Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDPI-21-006
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-01

CONDITIONS: Venous Reflux; Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GSV/SSV (Experimental): Incompetent Great and Small Saphenous Veins
  Interventions: Device: Venclose System (digiRF generator w EVSRF catheter)
- IPV (Experimental): Incompetent Perforator Veins
  Interventions: Device: Venclose MAVEN System (digiRF generator w MAVEN catheter)

INTERVENTIONS:
Device: Venclose System (digiRF generator w EVSRF catheter) — The Venclose System is intended for use in endovascular coagulation of blood vessels in patients with superficial vein reflux.
  Arms: GSV/SSV
Device: Venclose MAVEN System (digiRF generator w MAVEN catheter) — The Venclose MAVEN System is intended for use in endovascular coagulation of blood vessels in patients with perforator or tributary vein reflux.
  Arms: IPV

SUMMARY:
A Post-Market, Multi-Center, Prospective, Interventional Study for Treatment of Chronic Venous Disease of the Great and Small Saphenous Veins and Incompetent Perforator Veins.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 18 and older
2. Subject has CEAP clinical class C2 and higher.
3. Has been diagnosed with refractory symptomatic disease attributable to the GSV/SSV or IPV to be treated.
4. GSV/SSV or IPV to be treated that has an outward flow reflux duration of ≥ 0.5 seconds immediately after release of manual distal compression with subject standing or in Reverse Trendelenburg.
5. For GSV/SSV cohort only: GSV/SSV to be treated in a leg that has a diameter ≥4.5 mm.
6. For IPV cohort only: no more than two IPVs to be treated in a leg that have a diameter of ≥ 3.5 mm.
7. For IPV only: IPVs must be located under a healed or active ulcer.
8. Is able to ambulate.
9. Is able to comprehend and has signed the Informed Consent Form (ICF) to participate in the study.
10. Is willing and able to comply with the Clinical Investigation Plan and follow-up schedule.

Exclusion Criteria:

1. Has had previous treatment for venous insufficiency in the same target vein.
2. Has venous insufficiency secondary to venous obstruction proximal to the intended treatment site.
3. Has thrombus in the vein segment to be treated.
4. Has untreated critical limb ischemia from peripheral arterial disease.
5. Is undergoing active anticoagulant therapy for acute Deep Vein Thrombosis or other conditions (e.g., warfarin, direct oral anticoagulant or low molecular weight heparin) or has a history of Deep Vein Thrombosis within the last 6 months or hypercoagulable state.
6. Subjects with known bleeding and/or clotting disorders.
7. Has ABI <0.8
8. Subject is pregnant or breastfeeding
9. For GSV/SSV only: has a BMI >35.
10. For SSV only: has refluxing small saphenous vein thigh extensions (ex. Giacomini vein).
11. Unable to ambulate, or restrictive ambulation.
12. Has had prior venous procedures in the study limb within the last 30 days (including thrombolysis, thrombectomy, stenting, ablation, phlebectomy, visual or foam sclerotherapy).
13. Has undergone or is expected to undergo any major surgery within 30 days prior to or following the study procedure.
14. Has a condition, judged by the treating physician, that may jeopardize the subject's well-being and/or confound the results or the soundness of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Occlusion | 1-Month
  Cumulative Incidence of Occlusion
DVT & PE Serious Adverse Events | 1-Month
  Cumulative Incidence of Device and Procedural Related Deep venous thrombosis & Pulmonary Embolism Serious Adverse Events

SECONDARY OUTCOMES:
revised Venous Clinical Severity Score (rVCSS) | Baseline, 1-Week (+/- 2 days), 1-Month (+7 days), 3-Month (+/- 14 days), 6-Month (+/- 14 days), and 12- and 24-Month (+/- 30 days) visits
  Distribution of rVCSS score
ChronIc Venous Insufficiency Questionnaire - 20 (CIVIQ-20) | Baseline, 1-Month (+7 days), 3-Month (+/- 14 days), 6-Month (+/- 14 days) and 12- and 24-Month (+/- 30 days) visits
  Distribution of CIVIQ-20 score
Clinical Etiological Anatomical Pathophysiological (CEAP) | Baseline, 1-Week (+/- 2 days), 1-Month (+7 days), 3-Month (+/- 14 days), 6-Month (+/- 14 days), and 12- and 24-Month (+/- 30 days) visits
  Distribution of CEAP clinical class
Visual Analog Scale for Pain (VAS) | Baseline, Day 1 Index Procedure, 1-Week (+/- 2 days), 1-Month (+ 7 days), and 3-Month (+/- 14 days) visits
  Distribution of VAS Pain score
Recanalization | 1-Month (+7 days), 3-Month (+/- 14 days), 6-Month (+/- 14 days) and 12-Month (+/- 14 days) visits
  Proportion of Recanalization of treated veins
Duration of Procedure | Day 1 Index Procedure visit
  Mean Duration of Procedure
Endovenous Heat Induced Thrombosis (2-4) | 1-Month (+7 days) visit
  Cumulative incidence of device and procedural related endovenous heat-induced thrombosis (EHIT) Types 2-4

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - ClinRe, Thornton, Colorado
  - Pacific Vascular Institute, Kailua, Hawaii
  - Eastlake Cardiovascular, Roseville, Michigan
  - Englewood Hospital, Englewood, New Jersey
  - Atrium Health, Charlotte, North Carolina
  - Christus Health, Tyler, Texas
  - ClinRe, Colonial Heights, Virginia

IPD SHARING:
Plan to Share IPD: No